CLINICAL TRIAL: NCT01189279
Title: Safety and Pharmacokinetics Study of New Formulation of Bimatoprost in Patients With Alopecia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192024-053
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-06

CONDITIONS: Alopecia; Alopecia, Androgenetic; Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: bimatoprost Formulation A (Experimental): bimatoprost Formulation A applied topically to the scalp once daily on Day 1 and Days 4-17.
  Interventions: Drug: bimatoprost Formulation A
- Part 1: bimatoprost Formulation B (Experimental): bimatoprost Formulation B applied topically to the scalp once daily on Day 1 and Days 4-17.
  Interventions: Drug: bimatoprost Formulation B
- Part 2: bimatoprost Formulation C (Experimental): bimatoprost Formulation C applied topically to the scalp once daily on Day 1 and Days 4-17.
  Interventions: Drug: bimatoprost Formulation C

INTERVENTIONS:
Drug: bimatoprost Formulation A — bimatoprost Formulation A applied topically to the scalp once daily on Day 1 and Days 4-17.
  Arms: Part 1: bimatoprost Formulation A
Drug: bimatoprost Formulation B — bimatoprost Formulation B applied topically to the scalp once daily on Day 1 and Days 4-17.
  Arms: Part 1: bimatoprost Formulation B
Drug: bimatoprost Formulation C — bimatoprost Formulation C applied topically to the scalp once daily on Day 1 and Days 4-17.
  Arms: Part 2: bimatoprost Formulation C

SUMMARY:
This study will investigate the safety, tolerability, and pharmacokinetics of new formulation of bimatoprost following topical application in patients with alopecia. Two formulations of bimatoprost will be investigated in Part 1 and a third formulation of bimatoprost will be investigated in Part 2. Part 2 will begin after Part 1 has completed.

ELIGIBILITY:
Inclusion Criteria:

* Males with moderate male-pattern baldness (androgenic alopecia)
* Females with moderate female pattern hair loss
* Non-smoker or smoker with at least 30 days abstinence from smoking/using nicotine-containing products

Exclusion Criteria:

* Any dermatological condition of the scalp other than androgenic alopecia (males) or female pattern hair loss (females)
* Use of bimatoprost or other prostaglandin analogs within 3 months
* Prior use of scalp hair growth treatment (eg, finasteride, minoxidil) within 6 months
* Any prior hair growth procedures (eg, hair transplant or laser)
* Blood donation or equivalent blood loss within 90 days
* History of alcohol or drug addiction

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1 of the study was double-blind, followed by Part 2 which was open-label. No patients enrolled in Part 1 were enrolled in Part 2 of the study.
Period: Overall Study
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Started | 14 | 14 | 14
Completed | 13 | 14 | 13
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Customized [Number; unit: Participants]
  <45 years | 5 | 4 | 8 | 17
  45 to 64 years | 9 | 10 | 6 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 21
  Male | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Level (Cmax) Following a Single Dose of Bimatoprost
Description: Cmax is the maximum plasma level following a single dose of bimatoprost. Plasma is the fluid portion of the blood in which the cells are suspended.
Time Frame: Day 1
Population: Per Protocol: all subjects with no major protocol deviations
Measure: Mean (Standard Deviation); unit: Picograms/Milliliter (pg/mL)
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Number analyzed (Participants) | 14 | 14 | 14
Picograms/Milliliter (pg/mL) | 0.552 (0.575) | 1.77 (1.11) | 5.58 (3.66)

2. Primary Outcome: Maximum Plasma Level (Cmax) Following Multiple Doses of Bimatoprost
Description: Cmax is the maximum plasma level following multiple doses of bimatoprost. Plasma is the fluid portion of the blood in which the cells are suspended.
Time Frame: 17 Days
Population: Per Protocol: all subjects with no major protocol deviations
Measure: Mean (Standard Deviation); unit: Picograms/Milliliter (pg/mL)
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Number analyzed (Participants) | 13 | 14 | 13
Picograms/Milliliter (pg/mL) | 1.26 (0.60) | 3.01 (1.66) | 10.1 (7.0)

3. Secondary Outcome: Percentage of Patients With Clinically Significant Electrocardiogram (ECG) Findings
Description: An ECG is a tracing of the heart's electrical activity over time in waves with points identified at P, Q, R, S, and T [measured in milliseconds (ms)], as well as the heart rate [measured in beats per minute (bpm)]. Clinically significant abnormal results include maximum post-treatment QTcB>500 ms, maximum post-treatment QTcF>500 ms, maximum post-treatment QT interval >500 ms, PR interval 25% increase from baseline and >200 ms, QRS interval 25% increase from baseline and >100 ms, heart rate 25% increase from baseline and >100 bpm, and heart rate 25% decrease from baseline and <50 bpm.
Time Frame: 17 Days
Population: Safety Population: all subjects who received at least 1 dose of study medication
Measure: Number; unit: Percentage of Patients
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Number analyzed (Participants) | 14 | 14 | 14
Percentage of Patients | 0.0 (20.238) | 0.0 (23.460) | 0.0 (19.667)

4. Secondary Outcome: Number of Patients With an at Least 1-Grade Severity Increase in Local Scalp Tolerability by Patient Assessment
Description: Local scalp tolerability by patient assessment is based on a 4-point scale (0=None, 1=Mild, 2=Moderate, and 3=Severe) for 3 symptoms (burning, itching, and stinging). An at least 1-grade increase from baseline at any timepoint indicates a worsening of symptoms.
Time Frame: Baseline, 20 Days
Population: Safety Population: all subjects who received at least 1 dose of study medication
Measure: Number; unit: Patients
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Number analyzed (Participants) | 14 | 14 | 14
Patients
  Burning | 0 | 0 | 0
  Itching | 1 | 0 | 1
  Stinging | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With an at Least 1-Grade Severity Increase in Local Scalp Tolerability by Dermatologist Assessment
Description: Local scalp tolerability by dermatologist assessment is based on a 4-point scale (0=None, 1=Mild, 2=Moderate, and 3=Severe) for 5 symptoms (dryness/scaling, edema, erythema, folliculitis, and pigmentation). An at least 1-grade increase at any timepoint from baseline indicates a worsening of symptoms.
Time Frame: Baseline, 20 Days
Population: Safety Population: all subjects who received at least 1 dose of study medication
Measure: Number; unit: Patients
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Number analyzed (Participants) | 14 | 14 | 14
Patients
  Dryness/Scaling | 0 | 1 | 0
  Edema | 0 | 0 | 0
  Erythema | 4 | 0 | 0
  Folliculitis | 1 | 0 | 0
  Pigmentation | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Part 1: Bimatoprost Formulation A | Part 1: Bimatoprost Formulation B | Part 2: Bimatoprost Formulation C
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 7/14 | 6/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Bimatoprost Formulation A (N=14) | Part 1: Bimatoprost Formulation B (N=14) | Part 2: Bimatoprost Formulation C (N=14)
Headache (Nervous system disorders) | 3 | 1 | 1
Feeling Hot (General disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Application Site Folliculitis (Infections and infestations) | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.